CLINICAL TRIAL: NCT02789007
Title: Effects of Parabolic Flight on Spatial Cognition and Hippocampal Plasticity
Acronym: HypoCampus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Collaborators: Novespace (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2015-A02014-45
Record Dates: First submitted 2016-04-21; First posted 2016-06-02 (Estimated); Last update posted 2022-02-15 (Actual); Status verified 2016-11

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- parabolic flight (Other): To evaluate Structural and functional changes, Cognitive performance, and specifically spatial cognition, Key neurotrophins...
  Interventions: Other: Assess the impact of parabolic flight

INTERVENTIONS:
Other: Assess the impact of parabolic flight — MRI testing will be performed using a 3T MRI facility in Bordeaux close to Novespace (CHU Pellegrin).
  Spatial cognition will be assessed using a battery of in-house virtual paradigms General cognitive performance testing will include a wide range of cognitive functions, and particularly executive control using the Cognition Battery Mental status will be assessed on a tablet computer using a visual analogue scale Vigilant attention will be determined using the 3-min Psychomotor Vigilance Test (PVT) Blood samples (5 mL per collection) will be collected prior to neuroimaging by venepuncture

SUMMARY:
The main objective of this experiment is to assess the impact of parabolic flight on (1) spatial memory and orientation, (2) the changes in brain structure and function, and particularly the hippocampal formation, and (3) biochemical markers of stress and neuroplasticity.

A preliminary study will be performed with the aims (1) to test during weightlessness hardware used to administer visuo-spatial testing and (2) to determine the optimal body posture for testing under microgravity conditions (i.e. body posture for which change in visuo-spatial testing induced by weightlessness is maximal).

The main criteria are:

* Structural and functional changes of brain evaluated by fMRI;
* Cognitive performance, and specifically spatial cognition using a series computer-based tasks.
* Key neurotrophins determined in venous blood samples The criteria used in the preliminary experiment is visuo-spatial performance evaluated with a computer-based test assessing spatial cognition.

The investigators hypothesize that hippocampal structure and function, and particularly the dentate gyrus, will be altered after parabolic flight compared to ground based controls. Specifically, the 3 tested hypotheses are:

* Parabolic flight induces changes in hippocampal structure;
* Weightlessness induces changes in cognitive performance, and specifically spatial cognition;
* There is a correlation between changes in hippocampal structure and changes in visuo-spatial memory performance.
* There is a correlation between changes in hippocampal structure and changes in key neurotrophins.

The hypothesis tested during the preliminary experiment is that body posture affects the changes in spatial cognition performance.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers (men or women)
* Aged from 18 to 67
* Affiliated to a Social Security system and, for non-French resident, holding a European Health Insurance Card (EHIC)
* Who accepted to take part in the study
* Who have given their written stated consent
* Who has passed a medical examination similar to a standard aviation medical examination for private pilot aptitude (JAR FCL3 Class 2 medical examination). There will be no additional test performed for subject selection.

Subjects will be staff member of the team or of other teams participating in the parabolic flight campaign.

Exclusion Criteria:

* Person who took part in a previous biomedical research protocol, of which exclusion period is not terminated
* Person with medical history of claustrophobia
* Person with contraindication to MRI
* Pregnant women

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-03; Primary Completion 2019-03 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
Structural and functional changes of brain | baseline
  evaluated by fMRI

SECONDARY OUTCOMES:
Spatial Cognitive performance | baseline
  using a series computer-based tasks
Key neurotrophins | baseline
  determined in venous blood samples
visuo-spatial performance | baseline
  evaluated with a computer-based test assessing spatial cognition.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre DP Denise, PhD, Principal Investigator — CHU CAEN
Locations (1):
- Caen CHU, Caen, France

IPD SHARING:
Plan to Share IPD: No